CLINICAL TRIAL: NCT00109291
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Sequential Dose Escalation Study of the Safety, Pharmacodynamics, and Pharmacokinetics of Single Intravenous Doses of Peginesatide in Patients With Chronic Kidney Disease Who Are Not on Dialysis and Who Have Not Had Prior Erythropoiesis Stimulating Agent (ESA) Treatment
Brief Title: Safety of Single Doses of Peginesatide in Patients With Chronic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow enrollment
Sponsor: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFX01-02; 2005-000125-35 (EudraCT Number)
Record Dates: First submitted 2005-04-27; First posted 2005-04-27 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Anemia; Chronic Kidney Disease; Chronic Renal Failure
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; dialysis; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — peginesatide; hematide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Single injection of placebo administered intravenously
  Interventions: Drug: Placebo
- Peginesatide 0.025 mg/kg (Experimental): Single peginesatide dose of 0.025 milligram per kilogram (mg/kg) administered intravenously.
  Interventions: Drug: peginesatide
- Peginesatide 0.05 mg/kg (Experimental): Single peginesatide dose of 0.05 mg/kg administered intravenously.
  Interventions: Drug: peginesatide
- Peginesatide 0.10 mg/kg (Experimental): Single peginesatide dose of 0.10 mg/kg administered intravenously.
  Interventions: Drug: peginesatide

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: peginesatide
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide 0.025 mg/kg; Peginesatide 0.05 mg/kg; Peginesatide 0.10 mg/kg

SUMMARY:
To evaluate the safety profile of single intravenous (IV) dose levels of peginesatide in participants with chronic kidney disease(CKD) not on dialysis.

DETAILED DESCRIPTION:
This was a Phase 2a, randomized, double-blind, placebo-controlled, sequential dose escalation study conducted at a single clinical center. The study was designed to evaluate up to 6 treatment cohorts of 9 participants with CKD not on dialysis in the first cohort and 5 participants in each subsequent cohort. In each treatment cohort, participants were randomly assigned to receive either a single dose of peginesatide (n=7 in the first cohort, n=4 in subsequent cohorts) or placebo (n=2 in the first cohort, n=1 in subsequent cohorts). Participants were followed for a minimum of 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is informed of the investigational nature of this study and has given written, witnessed informed consent in accordance with institutional, local, and national guidelines;
2. Males or females ≥ 18 and ≤ 75 years of age. Pre-menopausal females (with the exception of those who are surgically sterile) must have a negative pregnancy test at screening; those who are sexually active must practice an adequate form of contraception for at least 2 weeks prior to study start, and must be willing to continue contraception for at least 4 weeks after receiving study drug;
3. Chronic kidney disease stage 3 or 4 (glomerular filtration rate [GFR] of 15-60 milliliter per minute (mL/min) within 28 days prior to administration of study drug,) not requiring dialysis;
4. Two hemoglobin values of ≥ 9 grams per deciliter (g/dL) and ≤ 11 g/dL within 14 days prior to administration of study drug, with one of the values drawn within 7 days prior to administration of study drug;
5. One serum ferritin level ≥ 100 micrograms per liter (µg/L) and one transferrin saturation ≥ 20% within 28 days prior to administration of study drug;
6. One serum folate level above the lower limit of normal within 28 days prior to administration of study drug;
7. One vitamin B12 level above the lower limit of normal within 28 days prior to administration of study drug;
8. Weight ≥ 45 kg within 28 days prior to administration of study drug;
9. One white blood cell count ≥ 3.0 x 10^9/L within 28 days prior to administration of study drug; and
10. One platelet count ≥ 140 x 10^9/L and ≤ 500 x 10^9/L within 28 days prior to administration of study drug.

Exclusion Criteria:

1. Prior treatment with any erythropoiesis stimulating agent;
2. History of pure red cell aplasia;
3. Red blood cell transfusion within 3 months prior to study drug administration;
4. Hemoglobinopathy (e.g., homozygous sickle-cell disease, thalassemia of all types, etc.);
5. Hemolysis based on medical judgment;
6. Chronic, uncontrolled, or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.);
7. C Reactive Protein (CRP) greater than 30 mg/L within 14 days prior to administration of study drug;
8. Significant infection within 4 weeks prior to study drug administration, per Investigator's clinical judgment ;
9. Febrile illness within 7 days prior to administration of study drug;
10. Uncontrolled or symptomatic secondary hyperparathyroidism;
11. Poorly controlled hypertension within 4 weeks prior to study drug administration, per Investigator's clinical judgment (e.g. systolic ≥ 170mm Hg, diastolic ≥ 100 mm Hg on repeat readings);
12. Epileptic seizure in the 6 months prior to study drug administration;
13. Chronic congestive heart failure (New York Heart Association Class IV);
14. High likelihood of early withdrawal or interruption of the study (e.g., myocardial infarction, severe or unstable coronary artery disease, stroke, respiratory, autoimmune, neuropsychiatric, or neurological abnormalities, liver disease including active hepatitis B or C, active HIV disease, or any other clinically significant medical diseases or conditions within the past 6 months that may, in the Investigator's opinion, interfere with assessment or follow-up of the patient);
15. Malignancy (except non-melanoma skin cancer);
16. Life expectancy < 12 months;
17. Anticipated elective surgery during the study period;
18. Previous exposure to any investigational agent within 4 months prior to administration of study drug or planned receipt during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-03; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | 28 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 28 days
  Pharmacokinetic parameters including Cmax, AUC0-t, AUC0-∞, t½ß, Vd, Vss, and Cl
Pharmacodynamic parameters | 28 days
  Pharmacodynamic parameters including reticulocytes, hemoglobin, reticulocyte hemoglobin content, and serum measures of iron stores (e.g., serum ferritin, transferrin saturation, and transferrin receptor protein)

CONTACTS AND LOCATIONS:
Overall Officials: Affymax, Study Director — Affymax, Inc.
Locations (1):
- Research Facility, London, United Kingdom